CLINICAL TRIAL: NCT00006329
Title: Comparison of Two Methods of Parathyroidectomy for Primary Hyperparathyroidism
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: NCRR-M01RR00042-1660; M01RR000042 (NIH)
Record Dates: First submitted 2000-10-04; First posted 2000-10-05 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-11

CONDITIONS: Hyperparathyroidism
Keywords: Radionuclide imaging; Surgery
MeSH Terms: conditions — Hyperparathyroidism

INTERVENTIONS:
Procedure: Minimally invasive radioguided parathyroidectomy

SUMMARY:
Parathyroid glands are small endocrine glands that secrete a hormone which controls blood calcium levels. Primary hyperparathyroidism (PH) is a common disorder whereby one or more of these glands may enlarge and overproduce their hormone. Subsequently, the elevated blood calcium can cause many other symptoms and problems. The standard treatment is surgical removal of the gland(s) causing the disorder. The standard safe and effective operation has been the bilateral open parathyroid exploration (BOPE). A newer procedure using a radioactive compound that concentrates in the parathyroid glands allows a more limited operation to find and remove the causative gland [Minimally-Invasive Radioguided Parathyroidectomy (MIRP)]. The radiation exposure is minimal and safe. Although the operation may prove to be less expensive, it is not certain whether it is as effective or as safe as BOPE. This study serves to directly compare the costs, the effectiveness, and the safety associated with each type of operation. All patients (adolescents and older) with PH are candidates to participate. The participants will be randomly assigned to the MIRP group or the BOPE group independently of patient or physician preferences. MIRP patients will undergo a sestamibi nuclear medicine scan to attempt to localize the specific parathyroid gland causing the hyperparathyroidism and subsequently a limited operation under local anesthesia to remove the single gland. Parathyroid hormone levels will be measured during the operation to ensure that the patient has been cured. If not, the standard BOPE procedure will be completed. The total cost of the care will be tracked for each group. Careful testing for complications such as vocal cord dysfunction will be done. General Health status and pain levels will be measured before and after each operation. Patient satisfaction with the operation and care will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Elevated serum calcium concentration on at least 2 occasions; if the value is <11.0 mg/dL, it must have been present for at least 6 months; if the serum albumin concentration is not normal, the ionized calcium level will be measured and must be elevated.
* Nephrolithiasis or documented bone mineral density less than 2.5 Standard Deviations below age matched means.
* Elevated or non-suppressed serum intact parathyroid hormone level

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Univ. of Michigan Hosp, Dept. of Surgery, Ann Arbor, Michigan, United States